CLINICAL TRIAL: NCT07255378
Title: Use of Vasopressin in Septic Shock.
Brief Title: Use of Vassopresin in Septic Shock Prospective Multicenter Observational Study With Medication
Acronym: VASO-2024
Status: Recruiting | Type: Observational
Sponsor: Jamil Cedeño Mora (Other)
Collaborators: Fundación para la Investigación Biomédica del Hospital Gregorio Maranon (Other); Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor-Investigator, Jamil Cedeño Mora, Consultant in Intensive Care Medicine. Head of Hemodynamics in the Intensive Care Unit., Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: VASO-2024
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock
Keywords: Norepinephrine; Septic Shock; Dose Threshold; Intensive Care Unit; Arginine Vasopressin Initiation
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Usage of vasopressin (VAP) as a second-line vasopressor in septic shock patients. — A state-of-the-art line of research in septic shock management focuses on the potential use of a second vasopressor agent. Current efforts aim to determine which drug should be used and the optimal timing for its initiation. In line with this, the Surviving Sepsis Campaign 2021 clinical guide recommends considering vasopressin-arginine (VAP) as a second-line vasopressor when norepinephrine (NAD) doses exceed 0.25 µg/kg/min, although this suggestion is based on limited evidence and remains weak.

SUMMARY:
The aim of this observational study is to examine real-world clinical practice regarding the use of vasopressin as a second-line vasopressor in adult patients admitted to Intensive Care Units (ICUs) with septic shock.

The study focuses on critically ill adults (≥18 years) diagnosed with septic shock and treated with norepinephrine and vasopressin.

The main research questions are:

* Does early initiation of vasopressin-defined by the norepinephrine dose at the time of introduction-reduce mortality in patients with septic shock?
* What is the impact of vasopressin as a second vasopressor on renal function and the progression of organ dysfunction in septic shock patients?

Participants will:

* Be admitted to an ICU with a diagnosis of septic shock.
* Receive vasopressin as an adjunct to norepinephrine for hemodynamic support.
* Be monitored daily throughout their ICU stay, with data collected through a dedicated REDCap system.
* Have relevant clinical data pseudonymized and incorporated into the study database for statistical analysis.

ELIGIBILITY:
Eligible patients for this study must comply with the following requirements.

* ICU admission with a septic shock diagnosis.
* Age 18 years or above at ICU admission.
* Use of vasopressin as an adjunct of norepinephrine.

For the purposes of this study, septic shock is defined by full compliance with the following criteria.

* Sustained arterial hypotension or serum lactate above 2 mmol/L.
* Adequate but unsuccessful fluid resuscitation.
* Vasopressor usage to maintain a mean arterial pressure above 65 mmHg.
* Probable or proven infectious etiology.

Patients with some of the following conditions will be automatically excluded.

* Pregnancy.
* Ischemic cardiogenic shock.
* Acute intestinal ischemia.
* Readmission to the Intensive Care Unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU-admitted patients treated at Spanish public hospitals participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Prognostic impact, in terms of all-cause mortality, of early VAP initiation in patients with septic shock. | From patient ICU-admission to 30 days after or patient ICU-discharge.

SECONDARY OUTCOMES:
Impact of vasopressin usage as a second vasopressor on renal function. | From patient ICU-admission to 30 days after or patient ICU-discharge.
  Renal function will be assessed using the Kidney Disease: Improving Global Outcomes (KDIGO) criteria for acute kidney injury (AKI). KDIGO stages range from 0 (no AKI) to 3 (severe AKI), with higher stages indicating worse renal function. KDIGO classification will be recorded at 24, 48, and 72 hours after vasopressin initiation, as well as the highest stage reached during the entire ICU stay.
  In addition to KDIGO staging, the need for renal replacement therapy (RRT) during admission will also be recorded as an indicator of progression to kidney failure.
Impact of VAP use as a second vasopressor on the progression of organ dysfunction. | From patient ICU-admission to 30 days after or patient ICU-discharge.
  Organ dysfunction will be measured using the Sequential Organ Failure Assessment (SOFA) score, which ranges from 0 (no organ dysfunction) to 24 (severe multi-organ failure). Higher scores indicate worse outcomes. SOFA score will be recorded at 24, 48, and 72 hours after vasopressin initiation, as well as the maximum SOFA score obtained during the ICU stay.

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Consorci Sanitari de Terrassa, Terrassa, BARCELONA
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario La Princesa, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Doce de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario y Politécnico de La Fe, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, ZARAGOZA

IPD SHARING:
Plan to Share IPD: No
The study protocol agreed upon with the supervising authorities explicitly excludes the possibility of doing so.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT07255378/Prot_SAP_001.pdf